CLINICAL TRIAL: NCT06211673
Title: Psychiatric Phenotype Characterization of Individuals With FOXP1 Syndrome
Acronym: FOXP1-PP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231331; 2023-A01981-44 (Other: IDRCB Number)
Record Dates: First submitted 2024-01-09; First posted 2024-01-18 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: FOXP1 Syndrome
Keywords: FOXP1 syndrome; hyperactivity; attention disorder; psychotic symptoms; autistic symptoms; sensory peculiarities; anxiety symptoms; sleeping disturbances; behavioral issues; general psychopathology; adaptive skills; agitation
MeSH Terms: conditions — Spasm; Cognition Disorders; Anxiety Disorders; Parasomnias; Psychomotor Agitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients and legal representatives: Minors and adults, without age limit, presenting with FOXP1 syndrome due to a genetic anomaly affecting the FOXP1 gene that has been identified, who have sought consultation at Necker-Enfants Malades Hospital, with at least one of the legal guardians or the legal representative being francophone.
  Interventions: Other: Semi-structured interviews; Other: Heteroquestionnaires

INTERVENTIONS:
Other: Semi-structured interviews — 3 semi-structured interviews will be administered to the legal guardians or legal representative of the patient:
  * Vineland Adaptive Behavior Scales II (VABS-II): assessment of adaptive skills;
  * Kiddie-SADS-Lifetime Version (K-SADS-PL): assessment of general psychopathology;
  * Autism Diagnostic Interview-Revised (ADI-R): assessment of autistic symptoms. The K-SADS-PL will be administered directly to the participant provided the participant is of an equivalent age of at least 5 years 11 months for receptive language and expressive language on the VABS-II, with raw scores of 35 and 92, respectively.
Other: Heteroquestionnaires — 7 heteroquestionnaires assessing: Hyperactivity symptoms and behavioral disorders measured by the ABC Attention deficit/hyperactivity symptoms measured by the Conners 3 scale and the SAID-P Psychotic symptoms measured by the adapted GPS-ID Sensory peculiarities measured by the Sensory Profile 2 Anxiety symptoms measured by the ADAMS Sleep disorders measured by the SDSC For children, the questionnaires: ABC, Sensory Profile 2, ADAMS, SDSC will be completed collectively by the legal guardians, and the questionnaires: Conners 3, SAID-P, adapted GPS-ID will be independently completed by each legal guardian. The same for adult patients with possible second caregiver. The questionnaires Conners 3, SAID-P and adapted GPS-ID will be completed twice, with a 28-day interval, at the time of inclusion and then after the semi-structured interviews.
  Other Names: Aberrant Behavior Checklist (ABC); Conners 3 scale; Scale of Attention in Intellectual Disability -Parent version (SAID-P); Adapted Glasgow Psychosis Screening Tool (adapted GPS-ID); Sensory Profile 2; Anxiety, Depression and Mood Scale (ADAMS); Sleep Disturbance Scale for Children (SDSC)

SUMMARY:
FOXP1 syndrome is a rare genetic disorder with a variable phenotype, characterized somatically by facial dysmorphia, dysphagia, hypotonia, relative or real macrocephaly, which may be associated with cerebral, cardiac, urogenital and ocular malformations. Psychiatrically, the syndrome manifests as a global developmental delay, then as mild to severe intellectual development disorder, speech and language impairments, behavioral issues that may include autistic features, hyperactivity and emotional lability. Assessing a cohort of 17 patients with FOXP1 syndrome, Trelles et al (2021) reported a significant frequency of autistic spectrum disorders, attention deficit/hyperactivity disorder (ADHD), and anxiety disorders. They also noted the presence of repetitive behaviors in the majority of patients and sensory-seeking behaviors. However, within the patient population at the Child and Adolescent Psychiatry Department of Necker Enfants Malades Hospital, a significant prevalence of psychotic disorders was observed. Additionally, families reported ineffectiveness and poor tolerance of methylphenidate in these patients. Therefore, it appears crucial to further characterize the psychiatric phenotype of individuals with FOXP1 syndrome and explore the link between agitation and psychotic prodromes.

DETAILED DESCRIPTION:
FOXP1 syndrome is a rare genetic pathology disorder with a variable phenotype, characterized somatically by facial dysmorphia, dysphagia, hypotonia, relative to or real macrocephaly, which may be associated with cerebral, cardiac, urogenital and ocular malformations. Psychiatrically, the syndrome manifests as a global developmental delay, then as mild to severe intellectual development disorder, speech and language impairments, behavioral abnormalities issues that may include autistic features, hyperactivity and emotional lability. Nevertheless, the investigative team of the study noted within the population of patients with FOXP1 syndrome followed in the child and adolescent psychiatry department of the Necker Enfants Malades hospital a significant prevalence of psychotic disorders. Furthermore, families report a lack of effectiveness and poor tolerance of methylphenidate in these patients. Also, it seems important to continue the characterization of the psychiatric phenotype of patients with FOXP1 syndrome and to question the link between agitation and psychotic prodromes. Assessing a cohort of 17 patients with FOXP1 syndrome, Trelles et al (2021) reported a significant frequency of autistic spectrum disorders, attention deficit/hyperactivity disorder (ADHD), and anxiety disorders. They also noted the presence of repetitive behaviors in the majority of patients and sensory-seeking behaviors. However, within the patient population at the Child and Adolescent Psychiatry Department of Necker Enfants Malades Hospital, a significant prevalence of psychotic disorders was observed. Additionally, families reported ineffectiveness and poor tolerance of methylphenidate in these patients. Therefore, it appears crucial to further characterize the psychiatric phenotype of individuals with FOXP1 syndrome and explore the link between agitation and psychotic prodromes.

The different elements that will be assessed include:

* hyperactivity symptoms;
* attention disorder symptoms;
* psychotic symptoms;
* autistic symptoms;
* sensory peculiarities;
* anxiety symptoms;
* sleeping disturbances;
* behavioral issues;
* general psychopathology;
* adaptive skills. Furthermore, the study will seek to determine whether agitation falls within the scope ofADHD (Attention Deficit Disorder with/without Hyperactivity) or whether if it is part of a context of emerging psychotic symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* Minor or adult patient, without age limit, presenting with FOXP1 syndrome due to an identified genetic anomaly affecting the FOXP1 gene;
* Patient who has sought consultationat Necker-Enfants Malades hospital;
* Legal guardians of the minor patient or legal representative of the adult patient, and the minor or adult patient capable of providing consent to participate in the study, informed about the study and not objecting to participation in the study.

Exclusion Criteria:

* Non French-speaking legal guardians or legal representatives of the patient;
* Illiterate legal guardians or legal representatives of the patient.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Minor or adult patient of the Necker-Enfants Malades hospital, without age limit, presenting FOXP1 syndrome secondary to an identified genetic anomaly affecting the FOXP1 gene and the holders of parental authority and legal representatives of patients.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Hyperactivity symptoms | Day 0
  Hyperactivity symptoms measured by the Aberrant Behavior Checklist (ABC). ABC: Behavioral assessment scale for individuals aged 5 to 58 years, comprising five subdomains: irritability and agitation, lethargy and social withdrawal, stereotyped behaviors, hyperactivity and non-collaboration, inappropriate speech. Validated tool for individuals with intellectual development disorders and those with autism spectrum disorders.
Attention deficit/hyperactivity symptoms | Day 0 and 21
  Attention deficit/hyperactivity symptoms measured by the Conners 3 scale and the Scale of Attention in Intellectual Disability - Parent version (SAID-P).
  Conners 3 scale: Scale for evaluating symptoms of Attention Deficit Hyperactivity Disorder (ADHD), Conduct Disorder, and Oppositional Defiant Disorder in individuals aged 6 to 18 years.
  SAID-P: Scale for assessing symptoms of Attention Deficit Hyperactivity Disorder (ADHD) in children with intellectual development disorders. The scale is currently undergoing validation.
Psychotic symptoms | Day 0 and 21
  Psychotic symptoms measured by the adapted Glasgow Psychosis Screening Tool (adapted GPS-ID).
  Adapted GPS-ID: Screening scale for psychotic symptoms in children with intellectual development disorders, adapted from the Glasgow Psychosis Screening Tool for use in Adults with Intellectual Disabilities (GPS-ID). The adapted scale has not yet been validated.
Autistic symptoms | Day 21
  Autistic symptoms measured by the Autism Diagnostic Interview-Revised (ADI-R). ADI-R: Semi-structured interview used for the diagnosis of Autism Spectrum Disorder in individuals with a developmental age beyond 24 months. Four domains are assessed: qualitative abnormalities in reciprocal social interaction; qualitative abnormalities in communication; restricted, repetitive, and stereotyped behaviors; evident developmental abnormalities at or before 36 months.
Sensory peculiarities | Day 0
  Sensory peculiarities measured by the Sensory Profile 2. Sensory Profile 2: Scale for assessing sensory integration abilities in individuals aged 7 months to 14 years 11 months, aiming to highlight the reaction profile (seeking, avoidance, sensitivity, registration) across different sensory channels and identify sensory systems (auditory, visual, tactile, proprioceptive, kinesthetic, oral) that may contribute to or hinder daily functional performance.
Anxiety symptoms | Day 0
  Anxiety symptoms measured by the Anxiety, Depression and Mood Scale (ADAMS). ADAMS: Scale for assessing anxiety and depressive symptoms in individuals with intellectual development disorders. The psychometric properties of this tool have been established in subjects aged 10 to 79 years of chronological age with mild to profound intellectual development disorders.
Sleeping disturbances | Day 0
  Sleep disturbances measured by the Sleep Disturbance Scale for Children (SDSC). SDSC: Scale for assessing sleep disorders comprising 25 items distributed across five factors (trouble initiating or maintaining sleep, parasomnia, excessive daytime sleepiness, sleep-related breathing disorder, non-restorative sleep), with the French version validated for individuals aged 4 to 16 years.
Behavioral issues | Day 0
  Behavioral disorders measured by the Aberrant Behavior Checklist scale (ABC).
General psychopathology | Day 14 (and day 28 with participant if applicable)
  General psychopathology measured by the Kiddie-SADS Semi-Structured Interview - Lifetime Version (K-SADS-PL).
  K-SADS-PL: Semi-structured diagnostic interview used to assess psychiatric disorders based on DSM-5 criteria in individuals aged 6 to 18 years. The tool includes a screening interview and five additional supplements (addressing mood, psychotic, anxiety, neurodevelopmental, and eating/addictive disorders) that will be administered based on identified signs observed during the screening interview. The K-SADS-PL involves separate interviews with parents and the subject themselves.
Adaptive skills | Day 7
  Adaptive skills measured by the Vineland Semi-Structured Interview II (VABS-II).
  VABS-II: Semi-structured interview used to assess the level of autonomy and adaptive capabilities in the areas of communication, daily living skills, socialization (and motor skills for individuals under 7 years of chronological age). The tool is applicable across all age groups and has been validated in individuals with intellectual development disorders.

SECONDARY OUTCOMES:
Agitation | Day 0
  Agitation measured by the "hyperactivity" subdomain of the Aberrant Behavior Checklist (ABC).
Correlation between agitation and symptoms of attention deficit/hyperactivity disorder on the one hand, and psychotic symptoms on the other hand | Day 0
  Assessment of the correlation between agitation measured by the "hyperactivity" subdomain of the Aberrant Behavior Checklist and symptoms of attention deficit/hyperactivity disorder measured by the "hyperactivity" subdomain of the Conners 3, on one hand, and psychotic symptoms measured by the adapted Glasgow Psychosis Screening Tool, on the other hand.
Psychometric properties of the Scale of Attention in Intellectual Disability - Parent version (SAID-P) | 23 months
  Assessment of the preliminary psychometric properties of the Scale of Attention in Intellectual Disability - Parent version (SAID-P).
Psychometric properties of the adapted Glasgow Psychosis Screening Tool (adapted GPS-ID) | 23 months
  Assessment of the preliminary psychometric properties of the adapted Glasgow Psychosis Screening Tool (adapted GPS-ID).

CONTACTS AND LOCATIONS:
Overall Officials: Maryse Pagnier, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Pauline Chaste, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alenezi S, Alyahya A, Aldhalaan H. Autism Spectrum Disorder (ASD) and Attention Deficit Hyperactivity Disorder (ADHD) With Language Impairment Accompanied by Developmental Disability Caused by Forkhead Box Protein 1 (FOXP1) Exon Deletion: A Case Report. Cureus. 2021 Dec 22;13(12):e20595. doi: 10.7759/cureus.20595. eCollection 2021 Dec. PMID 35103171
- [Background] Bekheirnia MR, Bekheirnia N, Bainbridge MN, Gu S, Coban Akdemir ZH, Gambin T, Janzen NK, Jhangiani SN, Muzny DM, Michael M, Brewer ED, Elenberg E, Kale AS, Riley AA, Swartz SJ, Scott DA, Yang Y, Srivaths PR, Wenderfer SE, Bodurtha J, Applegate CD, Velinov M, Myers A, Borovik L, Craigen WJ, Hanchard NA, Rosenfeld JA, Lewis RA, Gonzales ET, Gibbs RA, Belmont JW, Roth DR, Eng C, Braun MC, Lupski JR, Lamb DJ. Whole-exome sequencing in the molecular diagnosis of individuals with congenital anomalies of the kidney and urinary tract and identification of a new causative gene. Genet Med. 2017 Apr;19(4):412-420. doi: 10.1038/gim.2016.131. Epub 2016 Sep 22. PMID 27657687
- [Background] Chang SW, Mislankar M, Misra C, Huang N, Dajusta DG, Harrison SM, McBride KL, Baker LA, Garg V. Genetic abnormalities in FOXP1 are associated with congenital heart defects. Hum Mutat. 2013 Sep;34(9):1226-30. doi: 10.1002/humu.22366. Epub 2013 Jul 11. PMID 23766104
- [Background] Hamdan FF, Daoud H, Rochefort D, Piton A, Gauthier J, Langlois M, Foomani G, Dobrzeniecka S, Krebs MO, Joober R, Lafreniere RG, Lacaille JC, Mottron L, Drapeau P, Beauchamp MH, Phillips MS, Fombonne E, Rouleau GA, Michaud JL. De novo mutations in FOXP1 in cases with intellectual disability, autism, and language impairment. Am J Hum Genet. 2010 Nov 12;87(5):671-8. doi: 10.1016/j.ajhg.2010.09.017. Epub 2010 Oct 14. PMID 20950788
- [Background] Horn D, Kapeller J, Rivera-Brugues N, Moog U, Lorenz-Depiereux B, Eck S, Hempel M, Wagenstaller J, Gawthrope A, Monaco AP, Bonin M, Riess O, Wohlleber E, Illig T, Bezzina CR, Franke A, Spranger S, Villavicencio-Lorini P, Seifert W, Rosenfeld J, Klopocki E, Rappold GA, Strom TM. Identification of FOXP1 deletions in three unrelated patients with mental retardation and significant speech and language deficits. Hum Mutat. 2010 Nov;31(11):E1851-60. doi: 10.1002/humu.21362. PMID 20848658
- [Background] Lozano R, Gbekie C, Siper PM, Srivastava S, Saland JM, Sethuram S, Tang L, Drapeau E, Frank Y, Buxbaum JD, Kolevzon A. FOXP1 syndrome: a review of the literature and practice parameters for medical assessment and monitoring. J Neurodev Disord. 2021 Apr 23;13(1):18. doi: 10.1186/s11689-021-09358-1. PMID 33892622
- [Background] Meerschaut I, Rochefort D, Revencu N, Petre J, Corsello C, Rouleau GA, Hamdan FF, Michaud JL, Morton J, Radley J, Ragge N, Garcia-Minaur S, Lapunzina P, Bralo MP, Mori MA, Moortgat S, Benoit V, Mary S, Bockaert N, Oostra A, Vanakker O, Velinov M, de Ravel TJ, Mekahli D, Sebat J, Vaux KK, DiDonato N, Hanson-Kahn AK, Hudgins L, Dallapiccola B, Novelli A, Tarani L, Andrieux J, Parker MJ, Neas K, Ceulemans B, Schoonjans AS, Prchalova D, Havlovicova M, Hancarova M, Budisteanu M, Dheedene A, Menten B, Dion PA, Lederer D, Callewaert B. FOXP1-related intellectual disability syndrome: a recognisable entity. J Med Genet. 2017 Sep;54(9):613-623. doi: 10.1136/jmedgenet-2017-104579. Epub 2017 Jul 22. PMID 28735298
- [Background] O'Roak BJ, Deriziotis P, Lee C, Vives L, Schwartz JJ, Girirajan S, Karakoc E, Mackenzie AP, Ng SB, Baker C, Rieder MJ, Nickerson DA, Bernier R, Fisher SE, Shendure J, Eichler EE. Exome sequencing in sporadic autism spectrum disorders identifies severe de novo mutations. Nat Genet. 2011 Jun;43(6):585-9. doi: 10.1038/ng.835. Epub 2011 May 15. PMID 21572417
- [Background] Siper PM, De Rubeis S, Trelles MDP, Durkin A, Di Marino D, Muratet F, Frank Y, Lozano R, Eichler EE, Kelly M, Beighley J, Gerdts J, Wallace AS, Mefford HC, Bernier RA, Kolevzon A, Buxbaum JD. Prospective investigation of FOXP1 syndrome. Mol Autism. 2017 Oct 24;8:57. doi: 10.1186/s13229-017-0172-6. eCollection 2017. PMID 29090079
- [Background] Talkowski ME, Rosenfeld JA, Blumenthal I, Pillalamarri V, Chiang C, Heilbut A, Ernst C, Hanscom C, Rossin E, Lindgren AM, Pereira S, Ruderfer D, Kirby A, Ripke S, Harris DJ, Lee JH, Ha K, Kim HG, Solomon BD, Gropman AL, Lucente D, Sims K, Ohsumi TK, Borowsky ML, Loranger S, Quade B, Lage K, Miles J, Wu BL, Shen Y, Neale B, Shaffer LG, Daly MJ, Morton CC, Gusella JF. Sequencing chromosomal abnormalities reveals neurodevelopmental loci that confer risk across diagnostic boundaries. Cell. 2012 Apr 27;149(3):525-37. doi: 10.1016/j.cell.2012.03.028. Epub 2012 Apr 19. PMID 22521361
- [Background] Trelles MP, Levy T, Lerman B, Siper P, Lozano R, Halpern D, Walker H, Zweifach J, Frank Y, Foss-Feig J, Kolevzon A, Buxbaum J. Individuals with FOXP1 syndrome present with a complex neurobehavioral profile with high rates of ADHD, anxiety, repetitive behaviors, and sensory symptoms. Mol Autism. 2021 Sep 29;12(1):61. doi: 10.1186/s13229-021-00469-z. PMID 34588003